CLINICAL TRIAL: NCT06382610
Title: Pharmacokinetics of Melatonin Administered in Oral, Lotion, and Bubble Bath Formulations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Redlands (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 2024-002
Record Dates: First submitted 2024-04-19; First posted 2024-04-24 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-04

CONDITIONS: Sleep
Keywords: melatonin; transdermal; oral; pharmacokinetics
MeSH Terms: interventions — Melatonin

STUDY DESIGN:
Intervention Model Description: Repeated measures crossover trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Oral tablet (Active Comparator): 3 mg Tablets (Nature Made). Participants will need to fast for 2 hours prior to consumption and 2 hours after consumption.
  Interventions: Dietary Supplement: Melatonin
- Lotion (Experimental): Dr. Teal's Sleep Lotion with Melatonin, Lavender, and Chamomile. 3 g lotion applied to one arm (without washing for at least 4 hours).
  Interventions: Dietary Supplement: Melatonin
- Bubble bath (Experimental): Dr. Teal's Sleep Bath with Melatonin, Lavender, and Chamomile. 40L warm tap water maintained between 36.5 - 40 degrees C (98 - 104 degrees F) and 2 ml bubble bath. Participants will soak their feet and legs in the cooler for 15 minutes and then dry off (without rinsing or washing for at least 4 hours).
  Interventions: Dietary Supplement: Melatonin

INTERVENTIONS:
Dietary Supplement: Melatonin — Melatonin will be administered in three different forms

SUMMARY:
Melatonin is a hormone that promotes sleep that is available without a prescription in the United States. In addition to oral supplements, melatonin can be purchased in the form of lotions and bubble baths with unknown dosage and no frequency or age recommendations. In this study, researchers will examine how quickly melatonin in lotion and bubble bath is absorbed compared to oral tablets, as well as how long the melatonin lasts in the body.

DETAILED DESCRIPTION:
Melatonin is a hormone that promotes sleep that is available without a prescription in the United States. In addition to oral supplements, melatonin can be purchased in the form of lotions and bubble baths with unknown dosage and no frequency or age recommendations. A previous study (unpublished) has shown that a small amount of an over-the-counter lotion increases salivary melatonin levels by up to 1000 fold, a startling amount. Researchers will characterize the time course of the absorption and metabolism of lotion- and bubble bath-based melatonin compared to oral tablets in healthy 18-22 year olds.

The peak level, time to peak level and half-life of melatonin will be compared between the administration routes using a within-person (repeated measures) design and saliva sampling over 48 hours. Participants can choose specific days to participate within a one-month window, with a maximum of four sampling periods. All participants will collect control saliva samples (no melatonin treatment) one night at 10 PM and 4 AM. Participants will be asked to have two treatments 1) oral melatonin and 2) either lotion melatonin or bubble-bath melatonin. Participants can indicate if they have a preference for lotion vs. bubble bath or if they are willing to undergo both lotion and bubble bath treatments (adding a fourth sampling period). Order will be randomized.

For the treatments, saliva sampling times are as follows: Prior to melatonin administration (10 AM), then 15 min, 30 min, 45 min, 60 min, 90 min, 2 hours, 3 hours, 4 hours, 6 hours, 8 hours, 12 hours (10 PM), 18 hours (4 AM), 24 hours, 36 hours, and 48 hours after administration. Samples will be frozen at the participant's home until returned to the researchers at a later date. Melatonin in saliva samples will be quantitated via Enzyme Linked Immunosorbent Assay.

ELIGIBILITY:
Inclusion Criteria:

* University of Redlands student

Exclusion Criteria:

* Allergies or sensitivities to scented lotions or bath products
* Pregnancy

Ages: 18 Years to 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2024-05-19 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Salivary melatonin level | from immediately prior to administration to 48 hours post administration
  assessed via ELISA

SECONDARY OUTCOMES:
Side effects | from immediately prior to administration to 48 hours post administration
  Frequency of headache, drowsiness, dizziness, skin irritation, vivid dreams, and nightmares

CONTACTS AND LOCATIONS:
Overall Officials: Lisa E Olson, Ph.D., Principal Investigator — University of Redlands
Locations (1):
- University of Redlands, Redlands, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Upload salivary melatonin levels and side effect frequencies (all collected IPD) to National Sleep Research Resource (https://sleepdata.org/)
Supporting Information: Study Protocol, ICF
Time Frame: After relevant publication. Data will remain at the National Sleep Research Resource following their policy for keeping records.
Access Criteria: According to the National Sleep Research Resource